CLINICAL TRIAL: NCT00849160
Title: Non-comparative, Opened Study, Evaluating in HIV-1 Infected Patients With Undetectable Viral Load, Treated by an Antiretroviral Combination Including a Protease Inhibitor Boosted With Ritonavir and Administered by Oral Route Twice a Day, the Substitutability of the Current Protease Inhibitor Regimen by the Association Darunavir/Ritonavir 800/100 mg Once a Day to Maintain the Viral Load Under the 50 Copies/ml Limit of Detection After 24 Weeks of Treatment.
Brief Title: Study of Protease Inhibitor Regimen Switch in HIV-1 Infected Patients With Undetectable Viral Load to Prove the Non-inferiority of Once Daily Dose Regimen Versus the Current Twice Daily Regimen to Maintain the Viral Load Under the Limit of Detection.
Acronym: RADAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre de Recherches et d'Etude sur la Pathologie Tropicale et le Sida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREPATS 001
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: HIV-1 Infection; HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Darunavir/r (Experimental)
  Interventions: Drug: darunavir

INTERVENTIONS:
Drug: darunavir — darunavir/r 800/100 mg once daily by oral route, 48 weeks of treatment

SUMMARY:
Darunavir boosted with ritonavir (darunavir/r) is a powerful protease inhibitor, able to reduce the viral load in patients infected with multi-resistant HIV strains; In vitro and in vivo studies have shown that the induction of resistance mutations in the protease gene is much more difficult with the association darunavir/r compared to the other ritonavir-boosted protease inhibitors (PI/r), testifying of a significantly higher genetic barrier to resistance. Moreover, the tolerance to darunavir is good, and the pharmacologic profile of this molecule allows a once daily administration with a 800/100 mg dose in patients infected with a wild HIV strain or with a slightly resistant to darunavir/r strain.

Thus, we propose to evaluate the efficacy of the darunavir/r association once daily as a substitute to a protease inhibitor regimen administered twice daily in patients with undetectable viral load receiving a tritherapy including a protease inhibitor administered twice daily.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients
* Treatment with an association of 3 molecules including two Nucleotidic Reverse Trasncriptase Inhibitors and a ritonavir-boosted protease inhibitor BID, unchanged for at least one month
* At least two documented undetectable viral loads (under 50 copies/ml) within the last 3 months
* Naiive from darunavir
* Free from any opportunistic infection
* Creatinin < 3N
* ASAT & ALAT < 5N
* Haemoglobin > 7 g/dl
* Platelets > 50 000/mm3
* Negative pregnancy test for women of childbearing potential and use of a mechanic contraceptive during sexual relationships
* Signed informed consent

Exclusion Criteria:

* HIV-2 infected patients
* Treatment different from the association described in the inclusion criteria (2 NRTIs + 1 PI/r BID)
* Patients with a documented problem of treatment compliance within the last 12 months
* Ongoing active treatment against any opportunistic infection or tuberculosis
* Any critic concomitant condition (alcohol consumption, fatigue) that may jeopardize treatment compliance and/olr tolerance, and interfere with the protocol compliance
* Any concomitant treatment that may potentialize or inhibit hepatic cyotchrome-based enzymes
* Patient already treated with darunavir
* Patient treated with tipranavir, enfuvirtide, raltegravir, etravirine, and/or maraviroc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-05; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Undetectable viral load ( < 50 copies/ml) | Week 24

SECONDARY OUTCOMES:
Proportion of patients with undetectable viral load under 50 copies/ml | All visits
Proportion of patients in the situation of virologic failure defined as a viral load higher than 50 copies/ml confirmed with a second examen at least two weeks later. | All visits
CD4 lymphocytes count and evolution | All visits
Lipids balance evolution | All visits
Treatment tolerance | All visits
Measure of the darunavir/r concentrations variability and correlation with the potential adverse events and/or virologic failures. | All visits
Spermatic viral load (sub-study concerning 15 patients) | Day 0 and Week 48
Pharmacologic sub-studies | All visits

CONTACTS AND LOCATIONS:
Overall Officials: Jade Ghosn, MD, Principal Investigator — Centre Hsopitalier Universitaire de Bicêtre; Christine Katlama, MD, Study Director — Groupe Hospitalier Pitié-Salpêtrière
Locations (5):
- France (5):
  - Centre Hospitalier Universitaire de Bicêtre - Service de Médecine Interne et Maladies Tropicales, Le Kremlin-Bicêtre
  - Groupe Hospitalier Pitié-Salpêtrière - Service de Médecine Interne, Paris
  - Groupe Hospitalier Pitié-Salpêtrière - Service des Maladies Infectieuses et Tropicales, Paris
  - Hôpital Necker Enfants Malades - Service des Maladies Infectieuses et Tropicales, Paris
  - Hôpital Tenon - Service des Maladies Infectieuses et Tropicales, Paris